CLINICAL TRIAL: NCT04109729
Title: A Phase IB Study of Nivolumab in Combination With Radium-223 in Men With Metastatic Castration Resistant Prostate Cancer
Brief Title: Study of Nivolumab in Combination w Radium-223 in Men w Metastatic Castration Resistant Prostate Cancer
Acronym: Rad2Nivo
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI126006
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Nivolumab; Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Intervention Model Description: This is a phase 1, open label, prospective, non-randomized single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Radium-223 kBq/kg IV every 4 weeks for up to 6 doses. Nivolumab 480 mg IV every 4 weeks for up to 2 years.
  Interventions: Drug: Nivolumab; Drug: Radium-223

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480mg IV every 4 weeks for up to 2 years
  Other Names: Opdivo
Drug: Radium-223 — Radium-223 55 kilobecquerel (kBq)/kg IV q4 weeks for 6 cycles total
  Other Names: Xofigo

SUMMARY:
This is a phase 1, open label, prospective, non-randomized single arm study combining Radium-223 with nivolumab in men with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
Drug combination rationale Radium-223 is a calcium-mimetic radiopharmaceutical that has been approved for treatment of metastatic prostate cancer. Accumulating in areas of high bone turnover, such as bony metastases, radium-223 emits high energy alpha radiation within a narrow range thereby limiting toxicity (12). A pivotal phase III trial among patients with mCRPC and symptomatic bony metastases led to the approval of radium-223 (13). When compared to placebo, treatment with radium-223 resulted in an improved overall survival (OS) (3.6 months, HR 0.70, 95% confidence interval (CI) 0.58 to 0.83). This benefit was accompanied by no clinically significant difference in grade 3-4 adverse events between the two arms other than cytopenias. Patients also experienced a significant improvement in quality of life measures (14) with radium-223 compared to placebo.

Immunotherapy is a promising area of research in many areas of oncology. However, only PROVENGE is currently approved in mCRPC, with ipilimumab, pembrolizumab, and nivolumab previously demonstrating limited clinical efficacy. Beer et al evaluated ipilimumab monotherapy versus placebo in asymptomatic or minimally symptomatic men with mCRPC (15). Patients could not have visceral metastatic disease or prior chemotherapy. There was no improvement in OS, the primary endpoint of this study, with ipilimumab over placebo. The median OS was 28.7 months (95% CI, 24.5 to 32.5 months) for ipilimumab versus 29.7 months (95% CI, 26.1 to 34.2 months) with placebo (HR 1.11; 95.87% CI, 0.88-1.39; P = .3667). There was suggestion of some clinical response with the ipilimumab arm demonstrating more prostate specific antigen (PSA) responses (23% vs 8%) and a longer median progression free survival (PFS) (5.6 months vs 3.8 months). de Bono reported on the clinical efficacy of single agent pembrolizumab in mCRPC patients (16). They evaluated clinical activity based on the disease control rate (DCR), defined as no disease progression (i.e. complete response (CR) + partial response (PR) + stable disease (SD)). Eleven percent of patients had DCR of 6 months or greater, median follow up less than 12 months at the time of the study reporting. 19% of patients experienced any degree of PSA decline and 11% of patients had a 50% reduction or greater to PSA as the best response to therapy. Topalian et al evaluated the early safety and antitumor activity of monotherapy nivolumab in the basket trial CA209-003. Of the 296 patients treated, 17 were patients with castration-resistant prostate cancer (CRPC). However, no objective responses (complete response or partial response) were seen in this patient population (17). Overall the response rate is modest, demonstrating some activity with immunotherapy but suggesting that combination therapy may be a more attractive approach.

Recently the results of a prospective clinical trial of ipilimumab (CTLA-4 antagonist) and nivolumab (PD-1 antagonist) combination was reported in metastatic castration-resistant prostate cancer (18). 79 patients were treated and included patients who had previously progressed on docetaxel (cohort 2) and those who were docetaxel naïve (cohort 1). The objective response rate was 10% and 26% respectively. This therapy led to a significant number of significant adverse events, with a grade 3-4 adverse event (AE) rate of 51% and 39% respectively. A separate prospective pilot clinical trial in patients with high-risk disease as defined by presence of androgen receptor (AR)-V7 expression was also recently reported. The objective response rate was 25% in men with RECIST measurable disease and a 13% PSA response rate was observed overall (19). These studies demonstrate the significant improvement in clinical activity of combination immunotherapy over single-agent treatment in patients with metastatic castration-resistant prostate cancer. Overall the responses are still low even with the combination of multiple checkpoint inhibitors.

Many intrinsic mechanisms of resistance may account for this relative lack of efficacy including minimal baseline immune infiltration within the tumor (20), presence of immunosuppressive cells such as myeloid derived suppressor cells within the tumor microenvironment (21), and low tumor mutation burden leading to a lack of significant antigenicity (22).

External beam radiation therapy (EBRT) has been shown in preclinical models to alter the tumor microenvironment and may work synergistically with PD-1 inhibition. EBRT plus PD-1 inhibition resulted in improved tumor control compared to either agent alone in murine models (23). Alteration to PD-1 expression has also been observed with radium-223, suggesting potential synergy of these two strategies (24). Promotion of antigen presentation and antigen spreading may account for some of the beneficial effects of this combination in addition to the observed immunomodulatory effects on T-lymphocyte populations (25). The combination of EBRT plus checkpoint inhibitors has demonstrated promising efficacy in some early phase clinical trials (26,27).

Kwon et al evaluated men with mCRPC who had progressed on docetaxel to receive radiation therapy to a bone metastasis followed by randomization to ipilimumab or placebo (28). The median OS was prolonged with ipilimumab (11.2 months vs 10.0 months). However, given high toxicity early with ipilimumab, the primary endpoint was not statistically significant (HR 0.85; 95% CI 0.72-1.00; p=0.053). This benefit was even more evident in patients with good risk disease (median OS 22.7 mo vs 15.8 mo; HR 0.62, 95% CI 0.45-0.86; p=0.0038). This suggests that radiation therapy may provide added benefit to immunotherapy compared to ipilimumab monotherapy, especially in patients with a more favorable biology such as in patients lacking visceral metastasis (29) as will be tested in this clinical trial of nivolumab plus radium-223.

T-regulatory cells (defined as Cluster of Differentiation 4 (CD4)+/FOXP3+ T-cells) are immune suppressive. A higher concentration in peripheral blood mononuclear cells (PBMCs) and tumor infiltrating lymphocytes has been shown to correlate with an increased risk of disease relapse in localized renal cell carcinoma (30). Additionally, it also is associated with a worse prognosis in patients with metastatic melanoma (31). CD8+ T-cells are cytotoxic to tumor cells. A high level of CD8+ T-cells has recently been associated with an increased response to immunotherapy in patients with metastatic renal cell carcinoma (32). Cluster of differentiation 8 (CD8)+ and CD4+/FOXP3+ T-cell concentrations are associated with overall prognosis in patients with metastatic melanoma (33). The concentration of CD8+ lymphocytes is low in patients with prostate cancer (34). Animal models suggest that the combination of radiation therapy and checkpoint inhibitors provides synergistic activity through the alteration of the tumor microenvironment with increased CD8+ T-lymphocytes (35).

Radium-223 may overcome some of these mechanisms of resistance to single-agent checkpoint inhibitor therapy though immunomodulatory effects of radiation therapy to the microenvironment in addition to direct cytotoxicity of tumor cells leading to increased antigen presentation. We hypothesize that radium-223 plus nivolumab will result in significant, favorable tumor microenvironment alterations leading to significant clinical activity in mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged ≥ 18 years.
* Histologically confirmed adenocarcinoma of the prostate.
* Diagnosis of metastatic, castration-resistant prostate cancer without evidence of visceral metastasis.
* Symptomatic bone metastasis as determined by the treating physician.
* Castrate levels of testosterone as defined as < 50 ng/dL.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * White blood cell count (WBC) ≥ 2000/mm3
    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 10g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) unless there is a known history of Gilbert's syndrome.
    * Aspartate aminotransferase (AST)(SGOT)/Alanine aminotransferase (ALT)(SGPT) ≤ 5 × institutional ULN
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
* Highly effective contraception throughout the study and for at least 6 months after last study treatment administration if the risk of conception exists.
* Recovery to baseline or ≤ Grade 1 CTCAE v 5.0 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy as determined by the treating physician.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo-or hyperthyroid disease or other autoimmune diseases in the opinion of the treating physician that is clinically insignificant or not requiring systemic immunosuppressive treatment are eligible.
* Current use of immunosuppressive medication at the time of study enrollment, EXCEPT for the following permitted steroids:

  * Intranasal, inhaled, topical steroids, eye drops or local steroid injection (eg, intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography (CT) scan premedication).
* Prior or concurrent malignancy (other than adenocarcinoma of the prostate).

  --Note: Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial as approved by the Principle Investigator.
* The subject has uncontrolled, significant intercurrent or recent illness that would preclude safe study participation.
* Clinically significant cardiovascular disease: myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class IIB) or a serious cardiac arrhythmia requiring medication.
* Known HIV infection with a detectable viral load at the time of screening.

  --Note: Patients on effective antiretroviral therapy with an undetectable viral load at the time of screening are eligible for this trial.
* Known chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with a detectable viral load.

  --Note: Patients with an undetectable HBV viral load are eligible. Patients with an undetectable HCV viral load are eligible.
* Live attenuated vaccinations within 4 weeks of the first dose of radium-223 and while on trial is prohibited.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.4.1. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
To assess the frequency of grade 3 or greater non-hematologic treatment-emergent adverse events when combining nivolumab with Radium-223 | From cycle one day one until cycle 3 day 28 (each cycle is 28 days) - approximately 12 weeks
  Frequency of adverse events (AEs) characterized by seriousness, severity (as defined by CTCAE, version 5.0), duration, and relationship to study therapy. An increase in the clinically significant, non-hematologic grade 3 or greater toxicities above that observed in the Checkmate-214 trial will be considered unacceptable.
To assess the ctDNA reduction after 6 weeks of nivolumab treatment. | From cycle one day one until cycle 4 day 15 (each cycle is 28 days) - approximately 14 weeks
  Hypothesis: At least 40% of subjects with metastatic castrate resistant prostate cancer will have a Circulating tumor DNA (ctDNA) reduction after 6 weeks of therapy with Nivolumab in combination with Radium-233.
  An exact binomial test will be used to test the proportion of subjects with a ctDNA reduction at one-sided alpha = 0.05. The null proportion will be equal to 20%. The proportion of subjects with ctDNA reduction and 95% exact binomial confidence interval will be reported.

SECONDARY OUTCOMES:
To assess PSA progression free survival defined by the Prostate Cancer Working Group 3 (PCWG3). | up to 24 months
  Measurement of clinical activity of nivolumab in combination with Radium-223 in study population.
To assess correlation of bone metabolism markers with clinical response. | From cycle one day one until cycle 4 day 15 (each cycle is 28 days) - approximately 14 weeks
  Measurement of clinical activity of nivolumab in combination with Radium-223 in study population.
To assess response rates by serum PSA (defined by proportion of patients obtaining a 50% PSA reduction and the proportion of patients obtaining a 90% PSA reduction). | up to 24 months
  Measurement of clinical activity of nivolumab in combination with Radium-223 in study population.
To assess time to first symptomatic skeletal related event (defined as symptomatic fracture, surgery or radiation to bone, or spinal cord compression). | up to 24 months
  Measurement of clinical activity of nivolumab in combination with Radium-223 in study population.
To assess radiographic progression-free survival as defined by the PCWG3 criteria. | up to 24 months
  Measurement of clinical activity of nivolumab in combination with Radium-223 in study population.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maughan, MD, PharmD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No